CLINICAL TRIAL: NCT07181499
Title: A Study Evaluating the Efficacy and Safety of Pemetrexed Combined With Platinum-Based Chemotherapy Followed by Befotertinib in Patients With Non-Small Cell Lung Cancer After Third-Generation EGFR TKI Resistance
Brief Title: Sequential Chemotherapy With Befotertinib in Non-Small Cell Lung Cancer (NSCLC) Patients With Resistance to Third-Generation EGFR-TKI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-BF-IV028
Record Dates: First submitted 2025-09-10; First posted 2025-09-18 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: NSCLC; Adjuvant Drug Therapy; EGFR
MeSH Terms: interventions — Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group 1 (Experimental): pemetrexed (500 mg/m2) and carboplatin (AUC 5), administered every 3 weeks. After 2 to 4 cycles, received Befotertinib (75-100 mg)
  Interventions: Drug: Befotertinib; Drug: Pemetrexed + Carboplatin

INTERVENTIONS:
Drug: Befotertinib — Befotertinib was administered orally at a starting dose of 75 mg per day for 21 days, which could be increased to 100 mg per day if grade 2 or higher thrombocytopenia or headache did not occur within 21 days, or maintained at the original dose (75 mg per day) if grade 2 or higher thrombocytopenia or headache occurred within 21 days.
Drug: Pemetrexed + Carboplatin — pemetrexed (500 mg/m²) and carboplatin (AUC 5), administered every 3 weeks, for a total of 2~4 cycles.

SUMMARY:
Non-small cell lung cancer (NSCLC) accounts for over 85% of lung cancers. Approximately 30-40% of East Asian adenocarcinoma patients harbor EGFR mutations. Third-generation EGFR-TKIs achieve a median PFS of about 20 months as first-line therapy, but resistance eventually develops. Studies like MARIPOSA-2 confirm that amivantamab combined with chemotherapy ± lazertinib or immunotherapy regimens (ivucitinib/sintilimab + bevacizumab + chemotherapy) can extend median PFS post-resistance from approximately 4 months to 6-8 months. As a third-generation TKI, befitinib has demonstrated PFS of 16-22 months in both first-line and post-T790M mutation settings. This study aims to further evaluate the feasibility and safety of "pemetrexed + carboplatin followed by befotertinib" for patients resistant to third-generation TKIs.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Histologically or cytologically confirmed advanced or metastatic non-squamous NSCLC; and prior resistance to third-generation EGFR TKIs, with EGFR-sensitive mutations confirmed via tissue or blood samples (defined as: 19 Del or 21 L858R);
3. Exclusion of small cell lung cancer (SCLC) or squamous cell carcinoma (SqCC) transformation, and known NSCLC with clear targetable mutations for targeted therapy, such as HER2, MET amplification (GCN ≥ 5), KRAS G12C mutation, BRAF V600E mutation, RET fusion mutation, ALK fusion mutation, NTRK fusion mutation, etc.;
4. ECOG performance status (PS) score of 0-2;
5. Life expectancy of at least 12 weeks;
6. Ability to swallow oral medications;
7. Adequate organ system function, defined as follows and determined based on investigator judgment:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 10⁹/L
   2. Platelets ≥ 100 x 10⁹/L;
   3. Hemoglobin ≥ 9 g/dL (≥ 90 g/L). Note: Blood transfusions are permitted to achieve the required hemoglobin level;
   4. Total bilirubin ≤ 1.5 times the upper limit of normal (ULN);
   5. If no liver metastases: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; if liver metastases present: ≤ 5 × ULN;
   6. Creatinine ≤1.5 × ULN. If ≥1.5 × ULN, patients remain eligible if the Cockcroft-Gault-calculated creatinine clearance ≥50 mL/min (0.83 mL/s);
8. Female subjects of childbearing potential must have a negative serum pregnancy test within 3 days prior to study drug initiation and agree to use a medically approved highly effective contraceptive method (e.g., intrauterine device, oral contraceptives, or condoms) during the study and for 3 months after the last study drug administration; Male subjects with female partners of childbearing potential must be surgically sterilized or agree to use an effective method of contraception during the study period and for 3 months after the last study dose.
9. Voluntarily agree and be capable of adhering to the trial and follow-up procedures.
10. Be able to understand the nature of the trial and complete the written informed consent form.

Exclusion Criteria:

1. Rare EGFR mutations;
2. Prior treatment with pemetrexed and platinum-based chemotherapy regimens;
3. Advanced and/or symptomatic brain metastases (measurable or non-measurable) and/or leptomeningeal metastases;
4. Active hepatitis B (serum HBV DNA ≥10⁴ copies/mL [i.e., 20,000 IU/mL]), hepatitis C virus antibody positive, HIV antibody positive, or treponema pallidum antibody positive;
5. Women of childbearing potential with a positive serum pregnancy test within 7 days prior to treatment initiation, pregnant or lactating women, or male and female subjects not using effective contraception or planning pregnancy during treatment and for 3 months post-treatment;
6. Patients who used or require concomitant use of the following drugs within 14 days prior to the first dose or during treatment: drugs associated with QTc prolongation and/or risk of torsades de pointes ventricular tachycardia; strong CYP3A inhibitors or inducers;
7. Patients who underwent major surgery or immunotherapy within 4 weeks prior to the first dose; patients who received radiotherapy within 2 weeks prior to the first dose.
8. Imaging (CT or MRI) demonstrating tumor invasion of major vessels, or a high likelihood of tumor invasion into critical vessels causing fatal hemorrhage during the study period;
9. History of interstitial lung disease, drug-induced interstitial disease, or any clinically evident active interstitial lung disease; presence of idiopathic pulmonary fibrosis identified on baseline CT scan;
10. Other severe acute or chronic medical conditions, including uncontrolled diabetes, medical or psychiatric disorders, or laboratory abnormalities, that in the investigator's judgment may increase study-related risks or interfere with interpretation of study results;
11. Other conditions deemed by the investigator to be unsuitable for participation in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
progression free survival | From enrollment to the end of treatment at 12 months
  It refers to the time from the start of treatment until the tumor progresses or until death occurs for any reason (whichever occurs first).

SECONDARY OUTCOMES:
objective remission rate | From enrollment to the end of treatment at 12 month
  Objective Response Rate was defined as the percentage of participants whose tumor lesions disappear completely or diameters reduced by at least 30% as assessed by RECIST1.1.
Disease control rate | From enrollment to the end of treatment at 12 months
  Disease Control Rate was defined as the total percentage of participants except for those with tumor lesions diameters increased by at least 20% as assessed by RECIST1.1.
overall survival | From enrollment to the end of treatment at 36 months
  Overall survival was defined as the time from participants' treatment to their death due to any cause.
adverse event | From enrollment to the end of treatment at 12 months
  The number of participants with treatment-related adverse events as assessed by CTCAE v4.0 would be recorded and calculated after them participating into the study and taking the experimental drug.

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Pei, Study Director — The Fifth Affliated Hospital, Sun Yat-sen University; YingNi Lian, Principal Investigator — The First People's Hospital of Zhaoqing; DongYing Liu, Principal Investigator — Jiangmen Central Hospital; GuiNan Lin, Principal Investigator — Zhongshan People's Hospital, Guangdong, China; Shaodong Hong, Study Chair — Sun Yat-sen University
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The Cancer Center of The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong